CLINICAL TRIAL: NCT03176212
Title: Effect of Milk Fat Globule Membrane (MFGM) on Gut Barrier Protection in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Principal Investigator, Robert Ward, Associate Professor, Utah State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 101082
Record Dates: First submitted 2017-05-10; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Inflammation
Keywords: Gut permeability; Cytokine; Endotoxin
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beverage with milk fat globule membrane (Active Comparator): In this arm, subjects consumed a beverage
  Interventions: Dietary Supplement: Milk fat globule membrane
- Control (Placebo Comparator): In this arm, subjects consumed a beverage with identical macronutrients
  Interventions: Dietary Supplement: Milk fat globule membrane

INTERVENTIONS:
Dietary Supplement: Milk fat globule membrane

SUMMARY:
This study was designed to determine if an ingredient in milk fat can prevent gut leakiness induced by running at 80% maximum oxygen consumption (VO2max). In mouse studies, the milk fat ingredient, and individual components thereof, have been shown to reduce gut leakiness induced by intra peritoneal lipopolysaccharide (LPS) injections.

The investigators hypothesis is as follows: Compared to a sports drink with identical macro nutrient composition, a sports drink with milk fat globule membrane (MFGM) will reduce the change in gut leakiness induced by running at 90% VO2max for 30 minutes. The decrease in gut permeability change will be associated with a decreased area under the curve of plasma endotoxin for 5 hours following the exercise. In addition, decreased gut permeability will be associated with lower area under the curve values for inflammatory cytokines.

DETAILED DESCRIPTION:
A randomized, double-blind cross-over exercise trial was conducted with 14 runners on Utah State University campus. This population of 14 runners was selected from a larger population of 20 that was recruited to complete two initial trials. In two preliminary visits, the parameters necessary for conducting the experimental trial were determined. During the first visit, a baseline value was determined for gut permeability as well as aerobic capacity of runners. In the second visit the capacity to complete a run at 80% VO2max was tested and the effect of the exercise stress on gut permeability, plasma LPS and core temperature were measured.

Once a test population was selected, a randomized, double-blind, cross-over trial was conducted in which MFGM was tested for the ability to prevent a change in the exercise induced gut permeability.

During each testing session heart rate (HR), work output and core temperature (CT) were monitored. HR and CT were monitored by a CorTemp™ temperature pill which was ingested by the athletes prior to the trial (http://www.hqinc.net/pages/pill_page.html). In addition, blood was drawn at baseline (before depletion trial), immediately after the time trial, and again at 1h and 5h. Blood was analyzed for indices of training intensity (lactate), muscle damage (creatine kinase, cytokines), and gut barrier dysfunction (lipopolysaccharide, cytokines). In addition, immediately after the run athletes consumed a beverage with two carbohydrates (lactulose, and rhamnose). During the following six hours urine was collected and these sugars were measured via gas chromatography to determine the permeability of the gut.

Subject Recruitment Twenty, runners (ages 18-50) were initially recruited via campus flyers, advertisements in the local paper and weekly sports guide. Participants who had medical histories including: heart disease, uncontrolled hypertension, diabetes, Crohn's Disease, irritable bowel syndrome, colitis, Celiac disease, inflammatory or autoimmune diseases or lactose intolerance were excluded from the study. All subjects were instructed to avoid all anti-inflammatory medications for at least 24 h prior to any testing activity. On the morning of the first visit, approved subjects had body composition measured by BodPod (Life Measurement, Inc., Concord, CA). Participants were asked to refrain from any heavy exercise for 48 hrs before the first visit. Subjects were given a 50 ml tube containing the 5 g lactulose and 2 g rhamnose sugar probe and instructed to drink the probe 4hrs after they have finished breakfast to determine baseline gut permeability. Subjects were given a urine collection container and instructed to collect all urine for 6 hrs after ingestion of the probe. Subjects were not to eat lunch until 1.5 hrs after drinking the sugar probe. After 6 hrs of urine collection, subjects returned to the test site and performed a running VO2 max test.

Second Visit (approximately one week after first visit) Approximately 3 hrs after completion of breakfast, subjects reported to the test site to have blood drawn (to determine baseline plasma LPS), weight measured and to ingest a temperature probe. Participants started the exercise challenge (60 minute run at 80% VO2 max) approximately 4 hrs after completion of breakfast. The exercise challenge was conducted in a climate-controlled room at 22 °C without a fan. Subjects were monitored to ensure they were running at 80% VO2 max and were not allowed to consume water during the challenge. Immediately after the exercise challenge, participants consumed the sugar probes. Weight was measured, blood drawn (post-exercise plasma LPS) and subjects were instructed to collect their urine for the next six hrs. To facilitate re hydration and urine production, subjects were instructed to replace 150% of their fluid losses (pre to post exercise weight) by water intake.

After screening 20 subjects, a population of fifteen subjects agreed to participate in the cross-over trial. One subject dropped out due to a pregnancy, and four subjects could participate due to scheduling conflicts. One subject dropped out after sustaining a broken ankle that was not related to the study.

The third and fourth visits were the crossover portion of the experiment comparing MFGM to the vehicle. The 3rd and 4th visits were identical to the 2nd visit except participants drank either the fluid replacement vehicle or fluid replacement + MFGM 1 hr before the exercise challenge and again immediately following the exercise. Participants and personnel administering experimental protocols were blinded to treatments by use of coded, non-transparent drink containers. Subjects complete the 4th visit one week later and consume the vehicle beverage or the vehicle + MFGM.

For the crossover portion of the study, athletes were provided one of two beverages. The control beverage was formulated according to current sports nutrition guidelines for both pre- and post-workout nutrient delivery. It contained whey protein, sucrose, maltodextrins, chocolate flavoring and a small amount of butter oil. The test beverage was identical on a macro nutrient content, but contained a milk based ingredient called 'milk fat globule membrane.' This material is isolated from a byproduct of butter production, and is rich in phospholipids. The beverages were provided three hours prior to the exercise trial as well as immediately after. The test beverage contained a powder rich in MFGM that is produced by Arla Foods (Lacprodan PL-20) which contains roughly 20% phospholipids and 60% protein. In studies with mice, Dial et al have noted effects on gut protection in 1 h when animals are provided with phospholipids at 100mg/kg body weight. The second beverage was matched for macronutrient content, but did not contain the phospholipid powder.

Endpoints measured Change in gut Permeability To determine resting, baseline intestinal permeability the method of Pals was used. This method determines intestinal permeability by supplying the non-digestable sugars lactulose, and rhamnose and estimates intestinal and gastric permeability by recovery of these sugar probes in the urine. In healthy gut epithelia, lactulose has very limited transport across the gut barrier. Rhamnose crosses the small intestinal epithelia via a transcellular route and serves as internal control to account for gastric emptying rate, intestinal transit time and renal function. The larger lactulose molecule can only cross gut epithelia via a paracellular route through tight junctions. Therefore a higher ratio of lactulose to rhamnose recovered in the urine indicates compromised intestinal barrier function. Exercise stress has been demonstrated to significantly increase the urinary lactulose/rhamnose ratio . Similar to our proposed exercise stress model, this method has been used to demonstrate that running at 80% VO2max for an hour doubles gut permeability compared to baseline.

Change in plasma LPS: To assess endotoxemia, plasma LPS concentrations were measured via a kinetic activity as described by Nieman. Plasma LPS was measured from blood taken before exercise (baseline), immediately following, and at 1 and 5 hours after the exercise trial. Plasma LPS has been demonstrated to increase after endurance exercise bouts and is hypothesized to be the result of aberrant bacterial translocation of gut bacteria through compromised gut barrier. Elevated plasma LPS from baseline immediately after exercise has been demonstrated previously after a half-marathon, full marathon. It was anticipated that plasma LPS levels would increase after exercise stress and will be correlated to core body temperature and the lactulose/rhamnose index of gut barrier integrity.

Change in inflammatory Cytokines: Plasma levels of IL-6, TNFα, IL-10, IL-17, INFγ, IL-3, MCP-1, IL-15 and GMCSF were measured in the baseline and in the 1 h post exercise samples. Cytokine concentrations were determined by multiplex enzyme-linked immunosorbent assay (ELISA) by a commercial vendor (Quansys Biosystems, Logan, UT). These cytokines were selected based on a previous study investigating gut leakiness and MFGM consumption in an LPS-stimulated gut leakiness trial with mice. All cytokines were significantly upregulated in animals with leaky guts except GMCSF, and were significantly lowered in MFGM-fed animals compared to controls. Moreover, Ng et al demonstrated increased plasma levels of IL-10 and IL-6 (50% and 65.2% increase from baseline respectively) in runners immediately following a half marathon. Similarly, plasma levels of IL-6 and TNFα have been demonstrated to be increased from baseline immediately after a marathon. Based on the preliminary data and the aforementioned studies, it was anticipated that increased levels of inflammatory cytokines would be measured after the exercise challenge and it was hypothesized MFGM would abrogate this effect compared to the other recovery beverages.

Change in plasma creatine kinase: Creatine kinase was measured in samples taken before, immediately after and 1 hours after the exercise challenge. Creatine kinase was measured by using a commercial colorimetric kit (Sigma) in a 96-well UV/vis plate reader (Molecular Devices). Increased plasma creatine kinase is a well-established index of exercise induced muscle damage. In a similar study, cyclists riding at 85% VO2 max until exhaustion after glycogen depletion the previous day had less plasma creatine kinase when they consumed chocolate milk as a recovery drink compared to a carbohydrate replacement beverage.

Plasma Lactate: To assess anaerobic metabolism, plasma lactate will be measured at baseline, immediately after and 2 hours subsequent the exercise stress. Lactate will be measured using an enzymatic test kit (r-Biopharm, Marshall, MI).

The primary endpoint measured in this study was the lactulose/rhamnose ratios in urine and plasma LPS. The data were analyzed by single factor ANOVA and significant differences were explored with post-hoc testing. Core body temperature was measured in real time and was correlated with gut hypoxia and with gut leakiness.

All components measured in the blood (lactate, LPS, cytokines, and CK) were analyzed by a two factor ANOVA with time and treatment as variables. Lactate was included as it is generally considered to be an index of anaerobic activity. One other parameter were interested in is creatine kinase. As mentioned in the introduction, this enzyme is detected in the blood after intense exercise and is thought to correlate with damage to muscles. Furthermore, at least two studies with chocolate milk have noted that plasma CK is lower in athletes drinking chocolate milk vs. other recovery drinks.

Management plan All three PIs were actively involved in the planning and execution of this study, as well as in the sample processing and the analysis. Dr. Ward was responsible for formulation of the MFGM beverage. In addition, Dr. Ward was responsible for the GC-FID analysis of the urine. In addition, Dr. Ward will supervised a graduate student supported by this project.

Dr. Bressel recruited the athletes and helped with organizing the tests. In addition, Dr. Bressel supervised all of the performance trials and the collection of the exercise data.

Dr. Hintze was in charge of the blood and urine samples. The student (and perhaps Dr. Hintze) conducted the LPS the lactate and the CK assays. In addition, Dr. Hintze was responsible for proper sample handing of the blood and for the specimen delivery to Quansys Biosystems for the cytokine analysis.

All three PIs collaborated on the data analysis and on manuscript preparation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to run at 80%V02max for 30m, availability to complete the study.

Exclusion Criteria:

* Heart disease, uncontrolled hypertension, diabetes, Crohn's Disease, irritable bowel syndrome, colitis, celiac disease, inflammatory or autoimmune diseases, and lactose intolerance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in gut permeability via differential sugar test | Gut permeability was measured three times in this study. Once at baseline, and twice after the exercise challenges. The total time to complete the assessment was approximately 3 weeks.
  In this outcome, the barrier properties of the gut are assessed indirectly. Subjects consume a mixture of lactulose and mannitol. Mannitol is a monosaccharide and is passively absorbed from the gut and eliminated via the urine. Lactulose, on the other hand, is an indigestible disaccharide. If it appears in the urine, it is thought to pass into the body through loose tight junctions between the mouth and large intestine. If it reaches the large intestine, lactulose will be fermented by the microbiome.
  Subjects consume the sugar mixture and urine is collected for 6 hours. In this study, gut permeability was measured at baseline, and after after the running tests.

SECONDARY OUTCOMES:
Core temperature increase | This outcome was measured twice in a time frame of less than three weeks.
  Higher core temperatures are associated with increased gut permeability. Two of our primary measures were gut permeability assessments by the differential sugar test and plasma LPS. The increase in core temperature was included to give context to those measures. Prior to the exercise test, subjects consumed a thermometer pill and core temperature was monitored with a recording device.
Change in plasma lactate | This outcome was measured twice in a time frame of less than three weeks.
  Plasma lactate was measured as an index of exercise intensity. It was measured before the exercise challenge, and immediately after. It was also measured at 1 hour and 4 hours post exercise.
Change in plasma cytokines | This outcome was measured twice in a time frame of less than three weeks.
  To determine the systemic inflammatory response, plasma cytokines were measured before the exercise test and at 1h and 5h later. Plasma cytokines were measured with a multiplexed ELISA kit.
Change in plasma endotoxin | This outcome was measured twice in a time frame of less than three weeks.
  Higher levels of plasma endotoxin (aka LPS) are thought to occur due to a leaky gut
Change in plasma creatine kinase | This outcome was measured twice in a time frame of less than three weeks.
  Creatine kinase was measured as an index of muscle stress. It was measured before the exercise challenge, and immediately after. It was also measured at 1 hour and 4 hours post exercise.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dial EJ, Zayat M, Lopez-Storey M, Tran D, Lichtenberger L. Oral phosphatidylcholine preserves the gastrointestinal mucosal barrier during LPS-induced inflammation. Shock. 2008 Dec;30(6):729-33. doi: 10.1097/SHK.0b013e318173e8d4. PMID 18496240
- [Background] Pals KL, Chang RT, Ryan AJ, Gisolfi CV. Effect of running intensity on intestinal permeability. J Appl Physiol (1985). 1997 Feb;82(2):571-6. doi: 10.1152/jappl.1997.82.2.571. PMID 9049739
- [Background] Davis MS, Willard MD, Williamson KK, Steiner JM, Williams DA. Sustained strenuous exercise increases intestinal permeability in racing Alaskan sled dogs. J Vet Intern Med. 2005 Jan-Feb;19(1):34-9. doi: 10.1892/0891-6640(2005)192.0.co;2. PMID 15715045
- [Background] Lambert GP. Intestinal barrier dysfunction, endotoxemia, and gastrointestinal symptoms: the 'canary in the coal mine' during exercise-heat stress? Med Sport Sci. 2008;53:61-73. doi: 10.1159/000151550. PMID 19208999
- [Background] Smetanka RD, Lambert GP, Murray R, Eddy D, Horn M, Gisolfi CV. Intestinal permeability in runners in the 1996 Chicago marathon. Int J Sport Nutr. 1999 Dec;9(4):426-33. doi: 10.1123/ijsn.9.4.426. PMID 10660873
- [Background] Nieman DC, Henson DA, Dumke CL, Oley K, McAnulty SR, Davis JM, Murphy EA, Utter AC, Lind RH, McAnulty LS, Morrow JD. Ibuprofen use, endotoxemia, inflammation, and plasma cytokines during ultramarathon competition. Brain Behav Immun. 2006 Nov;20(6):578-84. doi: 10.1016/j.bbi.2006.02.001. Epub 2006 Mar 22. PMID 16554145
- [Background] Lambert GP, Lang J, Bull A, Pfeifer PC, Eckerson J, Moore G, Lanspa S, O'Brien J. Fluid restriction during running increases GI permeability. Int J Sports Med. 2008 Mar;29(3):194-8. doi: 10.1055/s-2007-965163. Epub 2007 Jul 5. PMID 17614027
- [Background] Ng QY, Lee KW, Byrne C, Ho TF, Lim CL. Plasma endotoxin and immune responses during a 21-km road race under a warm and humid environment. Ann Acad Med Singap. 2008 Apr;37(4):307-14. PMID 18461215
- [Background] Pritchett K, Bishop P, Pritchett R, Green M, Katica C. Acute effects of chocolate milk and a commercial recovery beverage on postexercise recovery indices and endurance cycling performance. Appl Physiol Nutr Metab. 2009 Dec;34(6):1017-22. doi: 10.1139/H09-104. PMID 20029509